CLINICAL TRIAL: NCT01204723
Title: Medications Development for the Treatment of Cannabis Related Disorders
Acronym: MTC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 14392; R01DA027131 (NIH)
Record Dates: First submitted 2010-09-14; First posted 2010-09-17 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Nicotine Withdrawal; Marijuana Dependence; Cannabis Dependence; Nicotine Dependence; Cannabis Abuse
Keywords: Marijuana Abuse; Nicotine Dependence; Nicotine Withdrawal; neurokinin Receptor; NK1 Receptor antagonist; Substance P; Recurrence; Substance Withdrawal Syndrome; Substance-Related Disorders; Disorders of Environmental Origin; Mental Disorders; Disease Attributes; Pathologic Processes; Tetrahydrocannabinol; Therapeutic Uses; Psychotropic Drugs; Analgesics, Non-Narcotic; Analgesics; Sensory System Agents; Peripheral Nervous System Agents; Neurotransmitter Agents; Molecular Mechanisms of Pharmacological Action; Narcotic Antagonists; cannabis
MeSH Terms: conditions — Marijuana Abuse; Tobacco Use Disorder; Recurrence; Substance Withdrawal Syndrome; Substance-Related Disorders; Disorders of Environmental Origin; Mental Disorders; Disease Attributes; Pathologic Processes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Behavioral Condition 1 (Experimental): Nicotine patch (21 mg) plus placebo oral cannabis (0 mg; 3 times a day on days 2-4, given once on day 5)
  Interventions: Drug: Placebo Aprepitant; Drug: Active Aprepitant
- Behavioral Condition 2 (Experimental): Placebo nicotine patch (0 mg) plus oral cannabis (10 mg, 3 times each day, days 2-4, day 5 given once)
  Interventions: Drug: Placebo Aprepitant; Drug: Active Aprepitant
- Behavioral Condition 3 (Experimental): Placebo nicotine patch (0 mg) plus placebo oral cannabis (0 mg, 3 times each day days 2-4, day 5 given once)
  Interventions: Drug: Placebo Aprepitant; Drug: Active Aprepitant

INTERVENTIONS:
Drug: Placebo Aprepitant — Placebo Aprepitant 0 mg once daily for 5 days
Drug: Active Aprepitant — Active Aprepitant 160 mg once daily for 5 days

SUMMARY:
The primary objective of this application is to test the neurobehavioral mechanisms and effects of aprepitant as a new cessation agent for cannabis, tobacco or both.

DETAILED DESCRIPTION:
Stress (emotional, physical, social) facilitates drug seeking behavior through the activation of the HPA axis, autonomic nervous system, and brain DA systems. Furthermore, alterations within several neuropeptide systems (CRF, Substance P, and others) also contribute to the role of stress in addiction. Central to this project is that anxiety and stress responses are modulated by substance P and its preferred target, the NK1 receptor. Therefore the aim of this pilot clinical trial is to determine the safety and efficacy of aprepitant (a neurokinin 1 (NK1) receptor antagonist). We hypothesize that the NK1 receptor antagonist, aprepitant, will be safe, tolerable and efficacious at reducing the withdrawal symptoms, cue craving, and reinforcement value for both cannabis and tobacco resulting from the cessation of either or both drugs. We will assess this hypothesis in the context of a carefully controlled human laboratory study in which subjects (N=72) will be randomized in a 3 x 2 factorial design to one of 3 behavioral conditions; a) withdrawn from both substances, b) withdrawn from tobacco only, or c) withdrawn from cannabis only, and to receive one of 2 medication dose conditions: placebo or aprepitant (160 mg/day). Medication will be administered for 5 days, followed by a cue challenge, choice procedure, and then a consequence (i.e., oral cannabis or a cigarette or money) also on day 5.

ELIGIBILITY:
Inclusion Criteria:

* Must meet DSM-IV/ICD-10 criteria for cannabis abuse or dependence
* Must be non-treatment seeking individuals
* Participant does not meet DSM-IV criteria for any current (i.e., criteria met at any point in the past 30 days) dependence on a substance other than alcohol, nicotine, caffeine, or marijuana or physiological dependence on alcohol requiring medical detoxification.
* No subjects who have trouble reading the English language or visual or hearing problems that may interfere with the collection of data
* Not currently taking other medications (with the exception of oral contraceptives) that would preclude safe participation in this study
* Must test negative for pregnancy prior to inclusion
* females using birth control pills must agree to use a condom during intercourse for 1 month after participation in study because the study medication will decrease the effectiveness of the birth control pill rendering it ineffective
* Should be in general good health
* No evidence of recent use of other illicit drugs on a urine toxicity screen prior to admission

Exclusion Criteria:

* Major current (within last 90 days) Axis I psychopathology (e.g., major depressive disorder, bipolar disorder, schizophrenia)
* Presence of significant medical illness (e.g., diabetes, cardiovascular disease, hypertension, cancer, epilepsy, kidney disease)
* Current, repeated illicit drug use (other than marijuana)
* Subject is breastfeeding or pregnant
* Concurrent therapy with drugs known to inhibit CYP3A4 activity
* Request for drug treatment
* Current parole or probation
* Recent history of significant violent or suicide behavior
* Allergic to sesame oil

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2009-08; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
withdrawal symptom severity, measured on a 0 (not at all) to 3 (severe) scale | collected on each study day
  Subjective experience of withdrawal symptoms for cannabis, tobacco, and both (eg: Irritability, Sleep difficulty, Chills, Nervousness)
"craving" measured using the Marijuana craving questionaire and the tobacco craving questionaire | collected on each study day
  Subjective measures of craving for cannabis, tobacco, and both Questionaires are anchored with strongly disagree to strongly agree (1-7)
reinforcing effects, as measured using the Multiple Choice Questionaire | collected each day of study
  Reinforcement value of cannabis and tobacco as measured by preference for money over the administration of either drug; questionaire has 70 questions and money value vs. drug ranges from 25 cents to 25 dollars 1-70.

SECONDARY OUTCOMES:
sleep quality | collected on each study day
  A VAS sleep questionnaire will be used each morning to assess daily sleep quality.
Neurocognitive Function | collected on days 1-4 of the study
  The purpose of examining the neurocognitive function of our participants on days 1-4 is to examine the safety of the co-administration of aprepitant at 160 mg/day with oral THC (dronabinol 10 mg) on brain function. Tasks used are the DSST - The Digit Symbol Substitution Test measures the learning of integrating visual and motor skills, and the SRTT- The Simple reaction Time Task is a well validated computerized test for assessing the effects of psychoactive drugs on performance.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | each day of study
  Blood pressure, pulse, and a Systematic Assessment For Treatment Emergent Events (SAFTEE) are collected daily. Electrocardiograms (EKGs) are collected at baseline and discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Haughey, Ph.D., Principal Investigator — University of Virginia School of Medicine, Dept. Psychiatry and Neurobehavioral Sciences
Locations (2):
- United States (2):
  - Clinical Pharmacological Research Unit (CPRU), University of Virginia School of Medicine, Charlottesville, Virginia
  - University of Virginia Center for Addiction Education and Treatment (UVA CARE), Charlottesville, Virginia

REFERENCES:
- [Derived] Gunderson EW, Haughey HM, Ait-Daoud N, Joshi AS, Hart CL. A survey of synthetic cannabinoid consumption by current cannabis users. Subst Abus. 2014;35(2):184-9. doi: 10.1080/08897077.2013.846288. PMID 24821356